CLINICAL TRIAL: NCT03671863
Title: Children Born With Club Feet: Ultrasound Diagnosis and Antenatal Assessment
Brief Title: Children Born With Club Feet
Acronym: CBCF
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0332
Record Dates: First submitted 2018-09-10; First posted 2018-09-14 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Clubfoot
Keywords: Ultrasound; Prenatal diagnosis; Congenital deformities; Perinatal outcome
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Infants who are treated for clubfoot: Infants who are treated for clubfoot in the reference reeducation center
  Interventions: Other: Invasive analysis (caryotype, CGH array); Other: Prenatal management

INTERVENTIONS:
Other: Invasive analysis (caryotype, CGH array) — Invasive analysis (caryotype, CGH array)
Other: Prenatal management — Prenatal management

SUMMARY:
Clubfoot is one of the most common birth defects, with a prevalence in Europe estimated between 1 and 4.5 for 1000 live birth.

It is useful to distinguish the forms of isolated clubfoot, and the forms related to others morphological abnormalities (complex clubfoot). For the complex forms, the clubfoot can be integrated in a syndromic association, be the consequence of a serious harm of the central nervous system, be associate to a genetic musculo-skeletal disease or wether be associated to a karyotype abnormality.

In those cases, the prognosis depends more about the associated morphological abnormalities that can be the beginning of a severe disability or incompatible with life or any anomaly of the karyotype that clubfoot itself.

In case of several morphological abnormalities, to propose invasive samples with realization of a karyotype and chromosome analysis with CGH array is a consensual attitude.

What the investigators should recommended to the parents in case of isolated form is less obvious and the question of antenatal investigations can not be answered clearly in the literature. Thus, the management of these patients may vary from one CPDP to another.

This study project will make it possible to analyze the management offered to patients whose fetuses have club feet and to study the results of the various examinations carried out in order to adapt the prenatal counselling and to define the best diagnostic strategy to propose to the future parents.

ELIGIBILITY:
Inclusion criteria:

* Congenital clubfoot uni or bilateral
* Have been treated in the reference center " Institut Saint Pierre, Plavas-les-flots, France "

Exclusion criteria:

- Non confirmed clubfoot after birth

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants with a clubfoot, antenatal diagned or not, treated at the " Institut Saint Pierre, Plavas-les-flots, France "
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Antenatal detection rate of clubfeet | At birth
  Antenatal detection rate of clubfeet in percentage

SECONDARY OUTCOMES:
Rate of isolated clubfoot among children followed for clubfoot | At birth
  Rate of isolated clubfoot among children followed for clubfoot in percentage
Rate of refered for second-degree examination | At birth
  Rate of refered for second-degree examination in percentage
Rate of invasive samples taken and their results | At birth
  Rate of invasive samples taken and their results in percentage
Rate of files submitted to our reference center committee | At birth
  Rate of files submitted to our reference center committee in percentage
Research rates of musculoskeletal genetic disease | At birth
  Research rates of musculoskeletal genetic disease in percentage
Rate of consultation with geneticist | At birth
  Rate of consultation with geneticist in percentage
Rate of consultation with a orthopedic surgeon | At birth
  Rate of consultation with a orthopedic surgeon in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Florent FUCHS, PhD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC